CLINICAL TRIAL: NCT04869566
Title: External Stressors Prior to Traumatic Knee Injury in Youth Athletes.
Status: Completed | Type: Observational
Sponsor: Linnaeus University (Other)
Responsible Party: Principal Investigator, Sofia Ryman Augustsson, Assiociate Professor, Linnaeus University
Other Study IDs: 2019-02609
Record Dates: First submitted 2021-04-28; First posted 2021-05-03 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Traumatic Knee Injury

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Athletes with traumatic knee injury: Youth athletes, aged 16-19, with traumatic knee injury

SUMMARY:
The aim of this study is to evaluate different aspects of mental stress aspects and its role as a potential risk factor for traumatic knee injury in youth athletes. Approximately 300 athletes (age 16-19) 50% women) who are involved in high risk sports (soccer, handball and floorball) will be included. The athletes will record his/hers traumatic knee injury together with information about training regimes and some details on injury mechanism on a web-based form. The form also includes questions about mental stressors, such as club exchange, changed game system in addition to conflict within and outside the family, etc, prior to injury.

The present study will contribute new knowledge on levels of muscle function and different aspects of mental stress factors that may be related to traumatic knee injury in young athletes.

ELIGIBILITY:
Inclusion Criteria:

Male and female sport high school athletes Aged 15-19 years Participating and competing in soccer, handball, or floorball

Exclusion Criteria:

Traumatic knee injury prior to sport high school.

-

Ages: 16 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Coaches of approximately 1400 athletes, aged 16-19 years, involved in sports related to high risk of knee injury (soccer, handball and floorball), at 70 high schools in Sweden, will be contacted and introduced to the study through email. The team coach at each school will distribute a web-based form to the athletes during their first, second or third year of the high-school period by email or through the school's intra-net system.
  We estimate that approximately 300 youth athletes (50% women) will be included. From the included participants, ahtletes with traumatic knee injury will be included for furhter analysis.
Sampling Method: Probability Sample
Enrollment: 329 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Number of participants that had occurred an injury during the last year | 12 months
  Data on injury are collected retrospectively using a web-designed (SurveyMonkey®) registration form.
Number of participants with one ore several mental stressors related to environmental and social conditions | 12 months
  Mental stressors, such as club exchange, changed game system, conflict within the family, examination at school etc will be recorded using a questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Sofia Ryman Augustsson, PhD, Principal Investigator — sofia.rymanaugustsson@lnu.se
Locations (1):
- Sofia Ryman Augustsson, Kalmar, Sweden

IPD SHARING:
Plan to Share IPD: No